CLINICAL TRIAL: NCT04505358
Title: A Randomized, Double-blind, Placebo-controlled Pilot Study to Evaluate the Biological Activity, Safety, and Pharmacokinetics of PU-AD in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Evaluate PU-AD in Subjects With Amyotrophic Lateral Sclerosis
Acronym: ALS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Samus Therapeutics company closure
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PU-AD-SD-0202
Record Dates: First submitted 2020-07-23; First posted 2020-08-10 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 3:2 randomization
Masking Description: Packages will be labeled to mask the distinction between PU AD and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 30 mg PU AD 3:2 ratio (Experimental): will be administered orally, as 30 mg active dose strength tablets qd on an empty stomach (1 hour prior to food or 2 hours after), at about the same time each day, via standard of care procedures at the site or at home. All subjects will have their first dose administered in clinic following completion of all baseline assessments
  Interventions: Drug: PU-AD
- 30 mg Placebo 3:2 ratio (Placebo Comparator): will be administered orally, as 30 mg placebo tablets (placebo has no active ingredients) qd on an empty stomach (1 hour prior to food or 2 hours after), at about the same time each day, via standard of care procedures at the site or at home. All subjects will have their first dose administered in clinic following completion of all baseline assessments
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PU-AD — active vs placebo
  Other Names: active
  Arms: 30 mg PU AD 3:2 ratio
Drug: Placebo — active vs placebo
  Other Names: non active
  Arms: 30 mg Placebo 3:2 ratio

SUMMARY:
This is a multicenter, Phase 2a, randomized, double-blind, placebo-controlled pilot study to assess the biological activity, safety and pharmacokinetics of PU-AD compared to placebo in ALS. It will be conducted in approximately 20 sites in the US. Approximately 30 subjects will be enrolled in this study; subjects will be randomized 3:2 to receive either PU-AD 30 mg or matching placebo qd, added onto any current stable background treatment.

DETAILED DESCRIPTION:
This is a multicenter, Phase 2a, randomized, double-blind, placebo-controlled pilot study to assess the biological activity, safety and pharmacokinetics of PU-AD compared to placebo in ALS. It will be conducted in approximately 20 sites in the US. Approximately 30 subjects will be enrolled in this study; subjects will be randomized 3:2 to receive either PU-AD 30 mg or matching placebo qd, added onto any current stable background treatment. Subjects who meet all inclusion criteria and none of the exclusion criteria will be eligible to participate in this study.

The study consists of a Screening Period (including background treatment stabilization, if required) (4 weeks), Treatment Period (24 weeks) and a safety Follow up Visit (4 weeks [±1 week] after the last dose of investigational medicinal product [IMP]). The expected study duration is up to 32 weeks.

The Screening visit will take place within 4 weeks prior to dosing, to assess eligibility of subjects. Eligible subjects will be randomized and then return to the site for baseline assessments at Week 1. During the 24 week Treatment Period, subjects will be administered 30 mg PU AD or matching placebo qd, orally, on an empty stomach (1 hour prior to food or 2 hours after), at about the same time each day.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ALS classified as Clinically Probable ALS or Clinically Definite ALS according to the El Escorial Revised Criteria4
2. ALS onset ≤ 18 months from Screening
3. Male or female aged 20 to 80 years old (inclusive)
4. ALSFRS-R ≥ 30
5. SVC ≥ 60% of predicted at Screening
6. Willing and able to provide informed consent
7. Concurrent medications riluzole and edaravone are permitted as long as the regimen is stable for at least 4 weeks prior to randomization and is expected to remain unchanged during the course of the study
8. Able to swallow tablets
9. Has been stable on medications that affect the CNS, for at least 4 weeks (including antidepressants, hypnotics and antipsychotics) and dose is not expected to change during the trial
10. Willing to abstain from benzodiazepine or other CNS depressant treatment for 24 hours prior to each clinic visit and night-time hypnotics for 8 hours prior to each clinic visit
11. Negative serum pregnancy test at Screening, for female subjects of childbearing potential
12. Male subjects:

Male subjects with female partners of childbearing potential are eligible to participate if they agree to ONE of the following methods of contraception from 21 days before the first dose of IMP through 4 months after the last dose of the IMP:

* Abstinence from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent
* Use of a male condom plus partner use of a contraceptive method with a failure rate of < 1% per year when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant.

In addition male subjects must refrain from donating sperm for the duration of the study and for 4 months after the last dose of the IMP.

Female subjects:

A female subject is eligible to participate if she is not pregnant and/or breastfeeding. Females of childbearing potential must agree to use a highly effective method of contraception consistently and correctly during the treatment period and for at least 3 months after the last dose of IMP.

Highly effective methods of contraception include, combined hormonal (estrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal, progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable, placement of an intrauterine device, placement of an intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner and true sexual abstinence, if it is the chosen life style of the subject.

Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only and the lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together

Exclusion Criteria:

1. Dependence on invasive or non-invasive mechanical ventilation (excluding continuous positive airway pressure for sleep apnea)
2. Has current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterological, respiratory, endocrinologic, neurologic (other than ALS), psychiatric, infectious, immunologic or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses of safety and pharmacologic effect in this study
3. Has a life expectancy of <1 years
4. Has had a history within the last 5 years of a serious infectious disease affecting the brain or head trauma resulting in protracted loss of consciousness
5. Has a history within the last 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ or in situ prostate cancer with a normal prostate specific antigen post treatment
6. Has a known history of human immunodeficiency virus, clinically significant multiple or severe drug allergies or severe post treatment hypersensitivity reactions
7. Has a "yes" answer to Columbia Suicide Severity Rating Scale (C-SSRS) suicidal ideation item 4 or 5, or any suicidal behavior assessment within 6 months of Screening, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening
8. Has a history of chronic alcohol or drug abuse/dependence within the past 5 years
9. Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening
10. History of bleeding disorder or predisposing conditions, blood clotting or clinically significant abnormal results on coagulation profile at Screening, as determined by the investigator
11. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV) or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening
12. Clinically significant 12 lead electrocardiogram (ECG) abnormalities, as determined by the investigator
13. Indication of impaired liver function as shown by an abnormal liver function profile at Screening (e.g., repeated values of aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≥ 2 × the upper limit of normal [ULN] and/or indication of impaired renal function at Screening) (e.g., repeated values of creatinine and blood urea nitrogen [BUN] ≥ 1.5 × ULN or estimated glomerular filtration rate [GFR] < 45 mL/minute/1.73 m2 and corroborating medical history and physical examination)
14. Any contraindications to lumbar puncture (LP), e.g., increased bleeding risk (platelet count < 100,000/µL, coagulopathies, anticoagulant drugs, antiplatelet therapy), lumbar spine deformity that might interfere with the procedure, evidence on magnetic resonance imaging (MRI) contraindicating LP, risk for cerebral herniation, space occupying lesion with mass effect, abnormal intracranial pressure due to increased CSF pressure, Arnold Chiari malformation, local infections at the puncture site and subject refusal of LP; abnormalities in the Screening CSF profile that are considered by the investigator to be clinically significant are exclusionary
15. Any major surgery or trauma within 12 weeks of Screening or during the Screening Period or any surgery planned during the study
16. Has active ocular condition, that in the opinion of the investigator, may alter visual acuity during the course of the study
17. Use of any drugs that are strong inhibitors of cytochrome (CYP) 450 (2D6 or 2C19) within 7 days or 5 half-lives of the inhibitor (whichever is longer), prior to administration of the first dose of IMP and/or plan to use throughout the study
18. Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives (if known) of the investigational drug, whichever is longer, prior to first dose of IMP in this study or is currently participating in another clinical study
19. Other unspecified reasons that, in the opinion of the investigator or Samus and/or its delegated medical monitor, place the subject at risk or make the subject unsuitable for the study or unable or unwilling to comply with the requirements of the study
20. Female subject of childbearing potential with positive pregnancy test or who is lactating
21. History or presence of conditions, which in the judgment of the investigator, are known to interfere with the absorption distribution, metabolism or excretion of drugs, such as prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy)
22. History of serious head injuries, unexplained syncope, loss of consciousness, CNS disease or dementia
23. Prior exposure to PU-AD or related compounds
24. Significant blood loss (> 450 mL) or has donated one or more units of blood or plasma within 6 weeks prior to study participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 12 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 24 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Slow Vital Capacity (SVC) | 12 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Slow Vital Capacity (SVC) | 24 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Handgrip strength using hand-held dynamometry | 12 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Handgrip strength using hand-held dynamometry | 24 weeks
  Clinical effect outcome assessments change from baseline (CFB)
6 Minute Walk Test (6MWT) | 12 weeks
  Clinical effect outcome assessments change from baseline (CFB)
6 Minute Walk Test (6MWT) | 24 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale (ROADS) | 12 weeks
  Clinical effect outcome assessments change from baseline (CFB)
Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale (ROADS) | 24 weeks
  Clinical effect outcome assessments change from baseline (CFB)

SECONDARY OUTCOMES:
Blood biomarkers (neurofilament light chain [NfL], phosphorylated neurofilament heavy chain [pNfH], Super oxide dismutase 1 (SOD1) | 12 weeks
  Biomarker change from baseline (CFB)
Blood biomarkers (neurofilament light chain [NfL], phosphorylated neurofilament heavy chain [pNfH], Super oxide dismutase 1 (SOD1) | 24 weeks
  Biomarker change from baseline (CFB)
CSF biomarkers (total tau [t-tau], phosphorylated tau231 [p-tau231], Neurofilament light chain (NfL), phosphorylated neurofilament heavy chain (pNfH), glial fibrillary acidic protein [GFAP], Transactive DNA binding protein 43 (TDP 43) | 12 weeks
  Biomarker change from baseline (CFB)
CSF biomarkers (total tau [t-tau], phosphorylated tau231 [p-tau231], NfL, pNfH, glial fibrillary acidic protein [GFAP], TDP 43 | 24 weeks
  Biomarker change from baseline (CFB)
Urinary biomarker (P75 extracellular domain [p75ECD]) | 12 weeks
  Biomarker change from baseline (CFB)
Urinary biomarker (P75 extracellular domain [p75ECD]) | 24 weeks
  Biomarker change from baseline (CFB)
Super oxide dismutase 1 (SOD1) (in subjects with known gene mutations: SOD1) in CSF and blood | 12 weeks
  Biomarker change from baseline (CFB)
Super oxide dismutase 1 (SOD1) (in subjects with known gene mutations: SOD1) in CSF and blood | 24 weeks
  Biomarker change from baseline (CFB)
Poly(GP) (in subjects with known gene mutations: Chromosome 9 open reading frame 72 (C9orf72) ) in CSF | 12 weeks
  Biomarker change from baseline (CFB)
Poly(GP) (in subjects with known gene mutations: Chromosome 9 open reading frame 72 (C9orf72) ) in CSF | 24 weeks
  Biomarker change from baseline (CFB)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, MD, Study Director — Samus Therapeutics Consultant

IPD SHARING:
Plan to Share IPD: No